CLINICAL TRIAL: NCT06409988
Title: External Validation of the SHA2PE Score and Its Comparison to the Oakland Score for the Prediction of Safe Discharge in Patients With Lower Gastrointestinal Bleeding
Brief Title: Safe Discharge in Lower Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Laura Gonzalez, Laura González González, Germans Trias i Pujol Hospital
Other Study IDs: EO ALTA SEGURA
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Lower GI Bleeding
Keywords: Discharge; lower gastrointestinal bleeding; Oakland score; SHA2PE score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lower gastrointestinal bleeding: Any >18 years old patient admitted to our hospital due to a lower gastrointestinal bleeding episode.
  Interventions: Other: Safe discharge

INTERVENTIONS:
Other: Safe discharge — There was no specific intervention, we only aimed to see if those admitted patients could have been safely dicharged from the emergency department.

SUMMARY:
The increasing incidence in lower gastrointestinal bleeding (LGIB) leads to a rise in hospital admission. Many LGBI are self-limiting thus the several scores to identify low risk patients suited to outpatient care have been described. We aim to compare two of this scores (Oakland score and SHA2PE score) in terms of performace to predict "safe discharge" from the emergency department.

DETAILED DESCRIPTION:
The growing incidence of lower gastrointestinal bleeding (LGIB) is leading to a rise in hospital admissions even though most LGIB episodes are self-limiting. The Oakland and SHA2PE scores were designed to identify patients best suited to outpatient care. Our aim is to validate the SHA2PE score and compare both of these scores in terms of predictiveness of safe discharge.

We conducted a retrospective observational study of LGIB patients admitted to our hospital between June 2014-June 2019. During this period, data from all LGIB episodes admitted from the ED were collected in an electronic anonymized database created specifically for this study. If any of the principal variables or critical information was missing, the patient was excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* All > 18 year old patients, male and women, admitted to our hospital between June 2014 and June 2019 because of LGIB (lower gastrointestinal bleeding).

Exclusion Criteria:

* Patients in whom LGIB occurred while already admitted for an other cause.
* Patients with LGIB transferred from another hospital due to comorbidities or severity of the gastrointestinal bleeding episode.
* Patients with post-polypectomy LGIB (endoscopic polypectomy <14 days before admission).
* Patients with gastrointestinal bleeding of unknown origin after a complete study.
* Patients who had undergone digestive tract surgery in the previous month.
* Patients with an ostomy.
* Patients with known colorectal cancer who had not undergone surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be selected after discharge from hospitalization in the gastroenterology department during the stablished time period.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Safe Discharge | After 1 month of follow-up from the hospital discharge
  Patients with lower gastrointestinal bleeding and absence of all the following: rebleeding, re-consulting for LGIB within 28 days after discharge, in-hospital mortality, requirement of red blood cell transfusion or endoscopic, radiological, or surgical haemostatic treatment.
Validation of SHA2PE score in our cohort | After 1 month of follow-up from the hospital discharge
  We aim to validate this score in a southern Europe cohort and compare it to the Oakland score

SECONDARY OUTCOMES:
Performance of Oakland score in safe discharge | After 1 month of follow-up from the hospital discharge
  We calculated the sensibility, specificity, positive and negative predictive values of the Oakland score in our patients cohort.
Performance of SHA2PE score in safe discharge | After 1 month of follow-up from the hospital discharge
  We calculated the sensibility, specificity, positive and negative predictive values of the SHA2PE score in our patients cohort.

OTHER OUTCOMES:
Demographic characterisctics of our cohort | After 1 month of follow-up from the hospital discharge
  Description of the main characteristics of the patients admitted due to lower gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: From July 2020 to January 2025
Access Criteria: The information will be shared under mail request, under a Word document if the IP of the study considers it necessary

REFERENCES:
- [Result] Oakland K, Chadwick G, East JE, Guy R, Humphries A, Jairath V, McPherson S, Metzner M, Morris AJ, Murphy MF, Tham T, Uberoi R, Veitch AM, Wheeler J, Regan C, Hoare J. Diagnosis and management of acute lower gastrointestinal bleeding: guidelines from the British Society of Gastroenterology. Gut. 2019 May;68(5):776-789. doi: 10.1136/gutjnl-2018-317807. Epub 2019 Feb 12. PMID 30792244
- [Result] Aoki T, Hirata Y, Yamada A, Koike K. Initial management for acute lower gastrointestinal bleeding. World J Gastroenterol. 2019 Jan 7;25(1):69-84. doi: 10.3748/wjg.v25.i1.69. PMID 30643359
- [Result] Lanas A, Garcia-Rodriguez LA, Polo-Tomas M, Ponce M, Alonso-Abreu I, Perez-Aisa MA, Perez-Gisbert J, Bujanda L, Castro M, Munoz M, Rodrigo L, Calvet X, Del-Pino D, Garcia S. Time trends and impact of upper and lower gastrointestinal bleeding and perforation in clinical practice. Am J Gastroenterol. 2009 Jul;104(7):1633-41. doi: 10.1038/ajg.2009.164. Epub 2009 May 5. PMID 19574968
- [Result] Lanas A, Garcia-Rodriguez LA, Polo-Tomas M, Ponce M, Quintero E, Perez-Aisa MA, Gisbert JP, Bujanda L, Castro M, Munoz M, Del-Pino MD, Garcia S, Calvet X. The changing face of hospitalisation due to gastrointestinal bleeding and perforation. Aliment Pharmacol Ther. 2011 Mar;33(5):585-91. doi: 10.1111/j.1365-2036.2010.04563.x. Epub 2011 Jan 5. PMID 21205256
- [Result] Oakland K. Changing epidemiology and etiology of upper and lower gastrointestinal bleeding. Best Pract Res Clin Gastroenterol. 2019 Oct-Dec;42-43:101610. doi: 10.1016/j.bpg.2019.04.003. Epub 2019 Apr 17. PMID 31785737
- [Result] Strate LL. Lower GI bleeding: epidemiology and diagnosis. Gastroenterol Clin North Am. 2005 Dec;34(4):643-64. doi: 10.1016/j.gtc.2005.08.007. PMID 16303575
- [Result] Chait MM. Lower gastrointestinal bleeding in the elderly. World J Gastrointest Endosc. 2010 May 16;2(5):147-54. doi: 10.4253/wjge.v2.i5.147. PMID 21160742
- [Result] Comay D, Marshall JK. Resource utilization for acute lower gastrointestinal hemorrhage: the Ontario GI bleed study. Can J Gastroenterol. 2002 Oct;16(10):677-82. doi: 10.1155/2002/156592. PMID 12420025
- [Result] Xavier SA, Machado FJ, Magalhaes JT, Cotter JB. Acute lower gastrointestinal bleeding: are STRATE and BLEED scores valid in clinical practice? Colorectal Dis. 2019 Mar;21(3):357-364. doi: 10.1111/codi.14529. Epub 2019 Jan 10. PMID 30537416
- [Result] Strate LL, Orav EJ, Syngal S. Early predictors of severity in acute lower intestinal tract bleeding. Arch Intern Med. 2003 Apr 14;163(7):838-43. doi: 10.1001/archinte.163.7.838. PMID 12695275
- [Result] Aoki T, Nagata N, Shimbo T, Niikura R, Sakurai T, Moriyasu S, Okubo H, Sekine K, Watanabe K, Yokoi C, Yanase M, Akiyama J, Mizokami M, Uemura N. Development and Validation of a Risk Scoring System for Severe Acute Lower Gastrointestinal Bleeding. Clin Gastroenterol Hepatol. 2016 Nov;14(11):1562-1570.e2. doi: 10.1016/j.cgh.2016.05.042. Epub 2016 Jun 14. PMID 27311620
- [Result] Kollef MH, O'Brien JD, Zuckerman GR, Shannon W. BLEED: a classification tool to predict outcomes in patients with acute upper and lower gastrointestinal hemorrhage. Crit Care Med. 1997 Jul;25(7):1125-32. doi: 10.1097/00003246-199707000-00011. PMID 9233736
- [Result] Oakland K, Jairath V, Uberoi R, Guy R, Ayaru L, Mortensen N, Murphy MF, Collins GS. Derivation and validation of a novel risk score for safe discharge after acute lower gastrointestinal bleeding: a modelling study. Lancet Gastroenterol Hepatol. 2017 Sep;2(9):635-643. doi: 10.1016/S2468-1253(17)30150-4. Epub 2017 Jun 23. PMID 28651935
- [Result] Oakland K, Kothiwale S, Forehand T, Jackson E, Bucknall C, Sey MSL, Singh S, Jairath V, Perlin J. External Validation of the Oakland Score to Assess Safe Hospital Discharge Among Adult Patients With Acute Lower Gastrointestinal Bleeding in the US. JAMA Netw Open. 2020 Jul 1;3(7):e209630. doi: 10.1001/jamanetworkopen.2020.9630. PMID 32633766
- [Result] Hreinsson JP, Sigurdardottir R, Lund SH, Bjornsson ES. The SHA2PE score: a new score for lower gastrointestinal bleeding that predicts low-risk of hospital-based intervention. Scand J Gastroenterol. 2018 Dec;53(12):1484-1489. doi: 10.1080/00365521.2018.1532019. Epub 2018 Nov 20. PMID 30457020